CLINICAL TRIAL: NCT02104661
Title: OxCarbazepine as a Neuroprotective Agent in MS: A Phase 2a Trial
Brief Title: Protective Role of Oxcarbazepine in Multiple Sclerosis
Acronym: PROXIMUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: National Multiple Sclerosis Society (Other); Novartis Pharmaceuticals (Industry); Barts & The London NHS Trust (Other); University College, London (Other); Royal Free Hospital NHS Foundation Trust (Other); Mid and South Essex NHS Foundation Trust (Other); St George's Healthcare NHS Trust (Other); Barnet and Chase Farm Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8722; 2013-002419-87 (EudraCT Number); 14-LO-0185 (Other: NRES Committee London - Harrow)
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Oxcarbazepine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OxCarbazepine Treatment (Experimental): Treated for 48 weeks with OxCarbazepine 150mg twice a day alongside current DMDs.
  Interventions: Drug: Oxcarbazepine
- OxCarbazepine Placebo (Placebo Comparator): Treated for 48 weeks with matched placebo 1 tablet twice a day alongside current DMDs
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxcarbazepine — Oxcarbazepine 150mg tablet, over encapsulated and back-filled with Microcrystalline Cellulose/Magnesium Stearate 1%.
  Other Names: Trileptal
  Arms: OxCarbazepine Treatment
Drug: Placebo — Placebo in a matched capsule containing Microcrystalline Cellulose/Magnesium Stearate 1%.
  Arms: OxCarbazepine Placebo

SUMMARY:
People with multiple sclerosis (MS) have nerve loss even without acute inflammatory relapses, as obvious in the progressive phase of disease. Drugs that may prevent nerve loss work better in earlier stages when it is difficult to measure progressive disability. But it is now possible to measure the nerve loss as neurofilament light (NFL) in the cerebrospinal fluid (CSF). This is a trial of a neuroprotective drug, oxcarbazepine, which showed benefit in an animal model of multiple sclerosis. The investigators will use an innovative outcome, a reduction in the content of NFL in the CSF, as well as the usual clinical disability and imaging methods, to measure the success of the oxcarbazepine as a neuroprotective agent in MS. The use of NFL, a surrogate marker of neurodegeneration, allows a blinded and accurate outcome.

DETAILED DESCRIPTION:
Patients who have been identified as potentially eligible for this trial and referred to us will be invited to take part in the study and provided with information given as a patient information sheet. This includes patients with clinical definite MS who are on any DMDs, have not had a MS relapses for at least 6 months and feel (subjective) or are observed (objective) to have progressing disability.

For screening patients will sign the informed consent form after discussion and make sure they fulfil inclusion and exclusion criteria, they will have a neurological and a brief suicidality assessment and will have safety blood and urine tests. Patients will have a lumbar puncture to measure NFL in CSF. If it is above the threshold, showing that there is ongoing damage to the myelin, we will invite them to continue in the trial.

Patients will have a baseline brain and spinal cord MRI and OCT, clinical/neurological examination and will have a repeat lumbar puncture and collection of blood, urine and saliva. Patients will be blindly randomised to oxcarbazepine vs placebo and given the bottles of medication with each participant's individualised label.

At two and four weeks after the baseline visit, patients will have a phone visit when investigators will collect details of new symptoms, new medication and generally advise participants. The tablets should have been increases to two tablets in the morning and two tablets in the evening.

Patients will be seen by the study team at 13 weeks after initiation of the drug and again at 25 and 37 weeks when they will have an OCT, lumbar puncture, collection of blood, urine and saliva after general, visual, neurological and cognitive assessments/questionnaires.

The final visit will be at week 48, when a final lumbar puncture, preceded by clinical measures including general, visual, neurological and cognitive assessments/questionnaires, MRI , OCT and blood, urine & saliva collection.

The measurement of NFL will be repeated from the CSF samples on the same at the end of the study to determine whether patients with MS who were on oxcarbazepine had a reduction in the levels of CSF NFL.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of definite multiple sclerosis
* Treatment with DMDs for at least 6 months prior to baseline visit*
* CSF NFL level ≥ 0.380ng/mL
* EDSS score between 3.5 and 6.0
* No history of relapses in the 6 months prior to the baseline visit
* A history of slow progression of disability, objective or subjective, over a period of at least 6 months prior to baseline
* Age 18-60 years

  * [Temporary interruption is permitted at the discretion of the investigator for a period of up to 8 weeks to prevent inflammatory MS reactivation. The cases where this could happen include for example switching DMDs that require a washout period as per clinical practice. When there are safety concerns, as in Lymphopenia or other side effects induced by the DMD, the interruption period can exceed 8 weeks as per clinical need. If reactivation of MS occurs with a relapse the investigator will assess if this meets withdrawal criteria 6.]

Exclusion Criteria:

* Pregnant or breastfeeding or unwilling to use adequate contraception.*
* Participants with a diagnosis of primary progressive PP MS or primary relapsing PR MS.
* A clinical relapse or pulsed intravenous or oral steroids in the 6 months preceding the baseline assessment.
* Participants presenting with medical disorder deemed severe or unstable by the CI such as poorly controlled diabetes or arterial hypertension, severe cardiac insufficiency, unstable ischemic heart disease, abnormal liver function tests (>2.5 times ULN) and abnormal complete blood count (in particular leukopenia, as defined by a lymphocyte count <500, neutrophil count <1.5 or platelet count <100, or thrombocytopenia <1.5 LLN), or any medical condition which, in the opinion of the investigator, would pose additional risk to the participant.
* Infection with hepatitis B or hepatitis C or human immunodeficiency virus.
* Exposure to any other investigational drug within 30 days of enrolment in the study.
* Judged clinically to have a suicidal risk in the opinion of the investigator based upon a clinical interview and the Columbia Suicide-Severity Rating Scale (CSSRS).
* Prior history of malignancy unless an exception is granted by the Investigator.
* History of uncontrolled drug or alcohol abuse within 6 months prior to screening.
* Past untoward reactions to OxCbz or Cbz
* Participants receiving OxCbz or Cbz in the previous 12 weeks from baseline

  * [Adequate methods of contraception are non hormonal methods such as barrier methods, intrauterine devices, surgical sterilisation (undergone by the participant or their partner). Female participants using hormonal only forms of contraception will be required to use an additional barrier method. True abstinence can be considered an acceptable method of contraception when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception. Non sexually active participants or those in same sex relationships will not be required to commence contraception.]

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Relative reduction of CSF neurofilament light chain levels | From baseline to week 48
  CSF obtained from lumbar punctures will be used to determine neurofilament light chain levels from baseline to 48 weeks between the active and placebo treated arms.

SECONDARY OUTCOMES:
Safety of Oxcarbazepine in multiple sclerosis patients | Ongoing throughout the trial
  Safety of OxCbz in multiple sclerosis patients as indicated by a comparison of adverse events to expected side effects outlined in the summary of product characteristics
Relative reduction of CSF neurofilament levels | baseline, 24 weeks and 48 weeks
  CSF obtained from lumbar punctures will be used to determine neurofilament light chain levels from baseline to 24 weeks and from 24 to 48 weeks between the active and placebo treated arms.
Change in clinical outcome measured by neurological examination. | Baseline, week 24 and week 48
  A neurological examination, including EDSS and Sloan chart will be performed by a study neurologist.
Change in clinical outcome measured by cognitive assessment | Baseline, week 12, 24, 36 and 48
  Cognitive assessment will consist of Symbol Digit Modalities Test (SDMT).
Change in patient reported outcomes measured by questionnaires | Baseline, weeks 12, 24, 36 and 48
  Patient questionnaires will include SF36, MSWS, MSIS-29 v2, Patient Pain Assessment and Patient Fatigue Assessment

OTHER OUTCOMES:
MRI scan to measure neurodegeneration | Baseline and week 48
  MRI scan will measure brain grey matter atrophy, spinal cord atrophy and three novel measures, that have potential to detect more specific neuroaxonal abnormalities and the effect on them of a sodium blocking channel agent, such as OxCbz: (i) total sodium concentration, (ii) axonal diameter and (iii) axonal density.
OCT to measure retinal nerve fibre layer (RNFL) for neurodegeneration | Baseline and weeks 24 and 48
  retinal nerve fibre layer (RNFL) constitutes a good surrogate marker of neurodegeneration of the unmyelinated axons in the optic nerve after optic neuritis it has also been demonstrated that RNFL thinning occurs in SPMS not previously affected by optic neuritis.
Biological samples collected to test for biomarkers of MS and correlation with response to OxCbz as a neuroprotector | Baseline, week 12, 24, 36 and 48
  These biomarkers of MS include immunological, viral, CNS components of cellular and genetic markers in CSF/serum/urine samples. We will use these to compare between people who are treated/respond to treatment with OxCbz

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Givannoni, Principal Investigator — Queen Mary University of London; Monica Calado Marta, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trapp BD, Peterson J, Ransohoff RM, Rudick R, Mork S, Bo L. Axonal transection in the lesions of multiple sclerosis. N Engl J Med. 1998 Jan 29;338(5):278-85. doi: 10.1056/NEJM199801293380502. PMID 9445407
- [Background] Leray E, Yaouanq J, Le Page E, Coustans M, Laplaud D, Oger J, Edan G. Evidence for a two-stage disability progression in multiple sclerosis. Brain. 2010 Jul;133(Pt 7):1900-13. doi: 10.1093/brain/awq076. Epub 2010 Apr 27. PMID 20423930
- [Background] Petzold A, de Boer JF, Schippling S, Vermersch P, Kardon R, Green A, Calabresi PA, Polman C. Optical coherence tomography in multiple sclerosis: a systematic review and meta-analysis. Lancet Neurol. 2010 Sep;9(9):921-32. doi: 10.1016/S1474-4422(10)70168-X. PMID 20723847
- [Background] Coles AJ, Cox A, Le Page E, Jones J, Trip SA, Deans J, Seaman S, Miller DH, Hale G, Waldmann H, Compston DA. The window of therapeutic opportunity in multiple sclerosis: evidence from monoclonal antibody therapy. J Neurol. 2006 Jan;253(1):98-108. doi: 10.1007/s00415-005-0934-5. Epub 2005 Jul 27. PMID 16044212
- [Background] Franklin RJ, Ffrench-Constant C. Remyelination in the CNS: from biology to therapy. Nat Rev Neurosci. 2008 Nov;9(11):839-55. doi: 10.1038/nrn2480. PMID 18931697
- [Background] Stys PK. General mechanisms of axonal damage and its prevention. J Neurol Sci. 2005 Jun 15;233(1-2):3-13. doi: 10.1016/j.jns.2005.03.031. PMID 15899499
- [Background] Barkhof F, Calabresi PA, Miller DH, Reingold SC. Imaging outcomes for neuroprotection and repair in multiple sclerosis trials. Nat Rev Neurol. 2009 May;5(5):256-66. doi: 10.1038/nrneurol.2009.41. PMID 19488083
- [Background] Altmann DR, Jasperse B, Barkhof F, Beckmann K, Filippi M, Kappos LD, Molyneux P, Polman CH, Pozzilli C, Thompson AJ, Wagner K, Yousry TA, Miller DH. Sample sizes for brain atrophy outcomes in trials for secondary progressive multiple sclerosis. Neurology. 2009 Feb 17;72(7):595-601. doi: 10.1212/01.wnl.0000335765.55346.fc. Epub 2008 Nov 12. PMID 19005170
- [Background] Kapoor R, Furby J, Hayton T, Smith KJ, Altmann DR, Brenner R, Chataway J, Hughes RA, Miller DH. Lamotrigine for neuroprotection in secondary progressive multiple sclerosis: a randomised, double-blind, placebo-controlled, parallel-group trial. Lancet Neurol. 2010 Jul;9(7):681-8. doi: 10.1016/S1474-4422(10)70131-9. Epub 2010 Jun 8. PMID 20621711
- [Background] Ebers GC, Heigenhauser L, Daumer M, Lederer C, Noseworthy JH. Disability as an outcome in MS clinical trials. Neurology. 2008 Aug 26;71(9):624-31. doi: 10.1212/01.wnl.0000313034.46883.16. Epub 2008 May 14. PMID 18480462
- [Background] Lycke JN, Karlsson JE, Andersen O, Rosengren LE. Neurofilament protein in cerebrospinal fluid: a potential marker of activity in multiple sclerosis. J Neurol Neurosurg Psychiatry. 1998 Mar;64(3):402-4. doi: 10.1136/jnnp.64.3.402. PMID 9527161
- [Background] Malmestrom C, Haghighi S, Rosengren L, Andersen O, Lycke J. Neurofilament light protein and glial fibrillary acidic protein as biological markers in MS. Neurology. 2003 Dec 23;61(12):1720-5. doi: 10.1212/01.wnl.0000098880.19793.b6. PMID 14694036
- [Background] Salzer J, Svenningsson A, Sundstrom P. Neurofilament light as a prognostic marker in multiple sclerosis. Mult Scler. 2010 Mar;16(3):287-92. doi: 10.1177/1352458509359725. Epub 2010 Jan 19. PMID 20086018
- [Background] Petzold A, Eikelenboom MJ, Keir G, Grant D, Lazeron RH, Polman CH, Uitdehaag BM, Thompson EJ, Giovannoni G. Axonal damage accumulates in the progressive phase of multiple sclerosis: three year follow up study. J Neurol Neurosurg Psychiatry. 2005 Feb;76(2):206-11. doi: 10.1136/jnnp.2004.043315. PMID 15654034
- [Background] Semra YK, Seidi OA, Sharief MK. Heightened intrathecal release of axonal cytoskeletal proteins in multiple sclerosis is associated with progressive disease and clinical disability. J Neuroimmunol. 2002 Jan;122(1-2):132-9. doi: 10.1016/s0165-5728(01)00455-6. PMID 11777552
- [Background] Petzold A, Baker D, Pryce G, Keir G, Thompson EJ, Giovannoni G. Quantification of neurodegeneration by measurement of brain-specific proteins. J Neuroimmunol. 2003 May;138(1-2):45-8. doi: 10.1016/s0165-5728(03)00092-4. PMID 12742652
- [Background] Norgren N, Rosengren L, Stigbrand T. Elevated neurofilament levels in neurological diseases. Brain Res. 2003 Oct 10;987(1):25-31. doi: 10.1016/s0006-8993(03)03219-0. PMID 14499942
- [Background] Kuhle J, Leppert D, Petzold A, Regeniter A, Schindler C, Mehling M, Anthony DC, Kappos L, Lindberg RL. Neurofilament heavy chain in CSF correlates with relapses and disability in multiple sclerosis. Neurology. 2011 Apr 5;76(14):1206-13. doi: 10.1212/WNL.0b013e31821432ff. Epub 2011 Feb 23. PMID 21346223
- [Background] Petzold A, Rejdak K, Plant GT. Axonal degeneration and inflammation in acute optic neuritis. J Neurol Neurosurg Psychiatry. 2004 Aug;75(8):1178-80. doi: 10.1136/jnnp.2003.017236. PMID 15258226
- [Background] Gunnarsson M, Malmestrom C, Axelsson M, Sundstrom P, Dahle C, Vrethem M, Olsson T, Piehl F, Norgren N, Rosengren L, Svenningsson A, Lycke J. Axonal damage in relapsing multiple sclerosis is markedly reduced by natalizumab. Ann Neurol. 2011 Jan;69(1):83-9. doi: 10.1002/ana.22247. Epub 2010 Dec 8. PMID 21280078
- [Background] Gnanapavan S, Grant D, Morant S, Furby J, Hayton T, Teunissen CE, Leoni V, Marta M, Brenner R, Palace J, Miller DH, Kapoor R, Giovannoni G. Biomarker report from the phase II lamotrigine trial in secondary progressive MS - neurofilament as a surrogate of disease progression. PLoS One. 2013 Aug 1;8(8):e70019. doi: 10.1371/journal.pone.0070019. Print 2013. PMID 23936370
- [Background] Al-Izki S et al. Selective targeting of neuroprotection to MS lesions: sodium channel blockers in experimental autoimmune encephalomyelitis. In: Multiple Sclerosis Journal.; 2011:S53-S276
- [Background] Koch MW, Polman SK. Oxcarbazepine versus carbamazepine monotherapy for partial onset seizures. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD006453. doi: 10.1002/14651858.CD006453.pub2. PMID 19821367
- [Background] May TW, Korn-Merker E, Rambeck B. Clinical pharmacokinetics of oxcarbazepine. Clin Pharmacokinet. 2003;42(12):1023-42. doi: 10.2165/00003088-200342120-00002. PMID 12959634
- [Background] Lidster K et al. Neuroprotection in a novel optic neuritis model. In: Multiple Sclerosis Journal.; 2011:S227-S505 17
- [Background] Solaro C, Restivo D, Mancardi GL, Tanganelli P. Oxcarbazepine for treating paroxysmal painful symptoms in multiple sclerosis: a pilot study. Neurol Sci. 2007 Jun;28(3):156-8. doi: 10.1007/s10072-007-0811-3. Epub 2007 Jun 30. PMID 17603770
- [Background] Lu CH, Kalmar B, Malaspina A, Greensmith L, Petzold A. A method to solubilise protein aggregates for immunoassay quantification which overcomes the neurofilament "hook" effect. J Neurosci Methods. 2011 Feb 15;195(2):143-50. doi: 10.1016/j.jneumeth.2010.11.026. Epub 2010 Dec 4. PMID 21134399
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Hobart J, Lamping D, Fitzpatrick R, Riazi A, Thompson A. The Multiple Sclerosis Impact Scale (MSIS-29): a new patient-based outcome measure. Brain. 2001 May;124(Pt 5):962-73. doi: 10.1093/brain/124.5.962. PMID 11335698
- [Background] Hobart J. The Multiple Sclerosis Impact Scale (MSIS-29). In: Quality of Life Measurement in Neurodegenerative and Related Conditions. Cambridge University Press; 2011:pp. 24-40
- [Background] Sumowski JF, Wylie GR, Deluca J, Chiaravalloti N. Intellectual enrichment is linked to cerebral efficiency in multiple sclerosis: functional magnetic resonance imaging evidence for cognitive reserve. Brain. 2010 Feb;133(Pt 2):362-74. doi: 10.1093/brain/awp307. Epub 2009 Dec 14. PMID 20008455
- [Background] Henderson AP, Trip SA, Schlottmann PG, Altmann DR, Garway-Heath DF, Plant GT, Miller DH. A preliminary longitudinal study of the retinal nerve fiber layer in progressive multiple sclerosis. J Neurol. 2010 Jul;257(7):1083-91. doi: 10.1007/s00415-010-5467-x. Epub 2010 Feb 9. PMID 20143110
- [Background] Black JA, Liu S, Carrithers M, Carrithers LM, Waxman SG. Exacerbation of experimental autoimmune encephalomyelitis after withdrawal of phenytoin and carbamazepine. Ann Neurol. 2007 Jul;62(1):21-33. doi: 10.1002/ana.21172. PMID 17654737
- [Background] Teunissen CE, Iacobaeus E, Khademi M, Brundin L, Norgren N, Koel-Simmelink MJ, Schepens M, Bouwman F, Twaalfhoven HA, Blom HJ, Jakobs C, Dijkstra CD. Combination of CSF N-acetylaspartate and neurofilaments in multiple sclerosis. Neurology. 2009 Apr 14;72(15):1322-9. doi: 10.1212/WNL.0b013e3181a0fe3f. PMID 19365053
- [Background] Fisniku LK, Chard DT, Jackson JS, Anderson VM, Altmann DR, Miszkiel KA, Thompson AJ, Miller DH. Gray matter atrophy is related to long-term disability in multiple sclerosis. Ann Neurol. 2008 Sep;64(3):247-54. doi: 10.1002/ana.21423. PMID 18570297
- [Background] Roosendaal SD, Bendfeldt K, Vrenken H, Polman CH, Borgwardt S, Radue EW, Kappos L, Pelletier D, Hauser SL, Matthews PM, Barkhof F, Geurts JJ. Grey matter volume in a large cohort of MS patients: relation to MRI parameters and disability. Mult Scler. 2011 Sep;17(9):1098-106. doi: 10.1177/1352458511404916. Epub 2011 May 17. PMID 21586487
- [Background] Furby J, Hayton T, Altmann D, Brenner R, Chataway J, Smith KJ, Miller DH, Kapoor R. A longitudinal study of MRI-detected atrophy in secondary progressive multiple sclerosis. J Neurol. 2010 Sep;257(9):1508-16. doi: 10.1007/s00415-010-5563-y. Epub 2010 May 1. PMID 20437181
- [Background] Chard DT, Jackson JS, Miller DH, Wheeler-Kingshott CA. Reducing the impact of white matter lesions on automated measures of brain gray and white matter volumes. J Magn Reson Imaging. 2010 Jul;32(1):223-8. doi: 10.1002/jmri.22214. PMID 20575080
- [Background] Rocca MA, Horsfield MA, Sala S, Copetti M, Valsasina P, Mesaros S, Martinelli V, Caputo D, Stosic-Opincal T, Drulovic J, Comi G, Filippi M. A multicenter assessment of cervical cord atrophy among MS clinical phenotypes. Neurology. 2011 Jun 14;76(24):2096-102. doi: 10.1212/WNL.0b013e31821f46b8. PMID 21670439
- [Background] Furby J, Hayton T, Anderson V, Altmann D, Brenner R, Chataway J, Hughes R, Smith K, Miller D, Kapoor R. Magnetic resonance imaging measures of brain and spinal cord atrophy correlate with clinical impairment in secondary progressive multiple sclerosis. Mult Scler. 2008 Sep;14(8):1068-75. doi: 10.1177/1352458508093617. Epub 2008 Jul 16. PMID 18632782
- [Background] Kalkers NF, Barkhof F, Bergers E, van Schijndel R, Polman CH. The effect of the neuroprotective agent riluzole on MRI parameters in primary progressive multiple sclerosis: a pilot study. Mult Scler. 2002 Dec;8(6):532-3. doi: 10.1191/1352458502ms849xx. PMID 12474997
- [Background] Horsfield MA, Sala S, Neema M, Absinta M, Bakshi A, Sormani MP, Rocca MA, Bakshi R, Filippi M. Rapid semi-automatic segmentation of the spinal cord from magnetic resonance images: application in multiple sclerosis. Neuroimage. 2010 Apr 1;50(2):446-55. doi: 10.1016/j.neuroimage.2009.12.121. Epub 2010 Jan 7. PMID 20060481
- [Background] Kearney H, Yiannakas MC, Abdel-Aziz K, Wheeler-Kingshott CA, Altmann DR, Ciccarelli O, Miller DH. Improved MRI quantification of spinal cord atrophy in multiple sclerosis. J Magn Reson Imaging. 2014 Mar;39(3):617-23. doi: 10.1002/jmri.24194. Epub 2013 Apr 30. PMID 23633384
- [Background] Inglese M, Madelin G, Oesingmann N, Babb JS, Wu W, Stoeckel B, Herbert J, Johnson G. Brain tissue sodium concentration in multiple sclerosis: a sodium imaging study at 3 tesla. Brain. 2010 Mar;133(Pt 3):847-57. doi: 10.1093/brain/awp334. Epub 2010 Jan 27. PMID 20110245
- [Background] Paling D et al. Total sodium concentration is increased in lesions and normal appearing white matter in Multiple Sclerosis. In: ISMRM.; 2012
- [Background] Schneider T, Wheeler-Kingshott CA, Alexander DC. In-vivo estimates of axonal characteristics using optimized diffusion MRI protocols for single fibre orientation. Med Image Comput Comput Assist Interv. 2010;13(Pt 1):623-30. doi: 10.1007/978-3-642-15705-9_76. PMID 20879283
- [Background] Schneider T. Mapping the axon diameter index in the corpus callosum is clinically feasible. In: ISMRM.; 2012
- [Background] Henderson AP, Trip SA, Schlottmann PG, Altmann DR, Garway-Heath DF, Plant GT, Miller DH. An investigation of the retinal nerve fibre layer in progressive multiple sclerosis using optical coherence tomography. Brain. 2008 Jan;131(Pt 1):277-87. doi: 10.1093/brain/awm285. Epub 2007 Dec 4. PMID 18056739
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Andersohn F, Schade R, Willich SN, Garbe E. Use of antiepileptic drugs in epilepsy and the risk of self-harm or suicidal behavior. Neurology. 2010 Jul 27;75(4):335-40. doi: 10.1212/WNL.0b013e3181ea157e. PMID 20660863
- [Background] Al-Izki S, Pryce G, Hankey DJ, Lidster K, von Kutzleben SM, Browne L, Clutterbuck L, Posada C, Edith Chan AW, Amor S, Perkins V, Gerritsen WH, Ummenthum K, Peferoen-Baert R, van der Valk P, Montoya A, Joel SP, Garthwaite J, Giovannoni G, Selwood DL, Baker D. Lesional-targeting of neuroprotection to the inflammatory penumbra in experimental multiple sclerosis. Brain. 2014 Jan;137(Pt 1):92-108. doi: 10.1093/brain/awt324. Epub 2013 Nov 27. PMID 24287115
- [Background] Davis A, Dobson R, Kaninia S, Espasandin M, Berg A, Giovannoni G, Schmierer K. Change practice now! Using atraumatic needles to prevent post lumbar puncture headache. Eur J Neurol. 2014 Feb;21(2):305-11. doi: 10.1111/ene.12307. Epub 2013 Dec 9. PMID 24320927
- [Background] Petzold A, Altintas A, Andreoni L, Bartos A, Berthele A, Blankenstein MA, Buee L, Castellazzi M, Cepok S, Comabella M, Constantinescu CS, Deisenhammer F, Deniz G, Erten G, Espino M, Fainardi E, Franciotta D, Freedman MS, Giedraitis V, Gilhus NE, Giovannoni G, Glabinski A, Grieb P, Hartung HP, Hemmer B, Herukka SK, Hintzen R, Ingelsson M, Jackson S, Jacobsen S, Jafari N, Jalosinski M, Jarius S, Kapaki E, Kieseier BC, Koel-Simmelink MJ, Kornhuber J, Kuhle J, Kurzepa J, Lalive PH, Lannfelt L, Lehmensiek V, Lewczuk P, Livrea P, Marnetto F, Martino D, Menge T, Norgren N, Papuc E, Paraskevas GP, Pirttila T, Rajda C, Rejdak K, Ricny J, Ripova D, Rosengren L, Ruggieri M, Schraen S, Shaw G, Sindic C, Siva A, Stigbrand T, Stonebridge I, Topcular B, Trojano M, Tumani H, Twaalfhoven HA, Vecsei L, Van Pesch V, Vanderstichele H, Vedeler C, Verbeek MM, Villar LM, Weissert R, Wildemann B, Yang C, Yao K, Teunissen CE. Neurofilament ELISA validation. J Immunol Methods. 2010 Jan 31;352(1-2):23-31. doi: 10.1016/j.jim.2009.09.014. Epub 2009 Oct 24. PMID 19857497